CLINICAL TRIAL: NCT00441935
Title: InterStim Prospective Database for Outcomes Research
Brief Title: InterStim Prospective Database
Status: Terminated | Type: Observational
Why Stopped: Shift in department's research interest
Sponsor: Kenneth Peters, MD (Other)
Collaborators: Corewell Health East (Other)
Responsible Party: Sponsor-Investigator, Kenneth Peters, MD, Principal Investigator, Corewell Health East
Organization: Corewell Health East (Other)
Other Study IDs: 2004-073
Record Dates: First submitted 2007-02-28; First posted 2007-03-01 (Estimated); Last update posted 2017-12-26 (Actual); Status verified 2017-12

CONDITIONS: Urinary Retention; Urinary Incontinence; Pelvic Pain
Keywords: Urinary Retention; Urinary Incontinence; Pelvic Pain
MeSH Terms: conditions — Urinary Retention; Urinary Incontinence; Pelvic Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Interstim Neuromodulation: Subjects undergoing implantation of an Interstim device for neuromodulation.
  Interventions: Device: Interstim Neuromodulation

INTERVENTIONS:
Device: Interstim Neuromodulation — Two stage procedure to implant an interstim device for neuromodulation.

SUMMARY:
The study is to collect information from patient charts and patient questionnaires to evaluate the effects of nerve stimulation therapy on urinary dysfunction.

DETAILED DESCRIPTION:
Men and women with urinary incontinence (leakage of urine), frequency, and bladder pain experience embarrassment, inconvenience, and a significant negative impact on their quality of life. Although traditional treatments such as medications, diet modification, and bladder training provide relief for some people, others do not experience improvement with these treatments. Recently, mechanical devices much like a heart pacemaker have been developed to stimulate the nerves (sacral and pudendal) responsible for controlling bladder function. During a two stage operation, a permanent electrical wire is implanted in the lower back and connected to a mechanical box (stimulator) implanted under the patients skin in the hip area.

Participants will be asked to complete a set of questionnaires (Intake Form, Urinary Incontinence Treatment Network (UITN) Sexual Activity Questionnaire, Interstitial Cystitis Symptom Index and Problem Index, voiding diary) within 60 days prior to the procedure. Preoperative clinical information such as primary diagnosis, history of failed therapies, and medical history will be collected from the physician office record, and operative information will be collected from the inpatient hospital record. After the two stage operation (3, 6, and 12 months, then yearly thereafter as long as the device is in place) participants will be sent questionnaires. Upon completion and return to the study site

ELIGIBILITY:
Inclusion Criteria:

* All patients at least 18 years of age scheduled for sacral nerve stimulator implantation at William Beaumont Hospital, Royal Oak, Michigan who give informed consent to participate in the project.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients at least 18 years of age scheduled for sacral nerve stimulator implantation at William Beaumont Hospital, Royal Oak
Sampling Method: Non-Probability Sample
Enrollment: 736 (Actual)
Dates: Start 2004-04; Primary Completion 2016-12-16 (Actual); Study Completion 2016-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Peters, MD, Principal Investigator — Corewell Health East
Locations (1):
- William Beaumont Hospital, Royal Oak, Michigan, United States